CLINICAL TRIAL: NCT06769841
Title: Parent-Related Factors Associated With Sleep in Young Children
Status: Active, not recruiting | Type: Observational
Sponsor: Marmara University (Other)
Collaborators: E-BEBEK Retail Joint Stock Company (Unknown)
Responsible Party: Sponsor
Other Study IDs: 09.2024.1086
Record Dates: First submitted 2025-01-06; First posted 2025-01-10 (Actual); Last update posted 2025-08-22 (Actual); Status verified 2025-06

CONDITIONS: Child Sleep; Parenting; Parent-child Relations
Keywords: sleep; parent; infant

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
Sleep plays a crucial role in supporting a child's healthy development, growth, and overall well-being. While many children develop healthy sleep patterns, 20-30% of infants experience sleep problems. Beyond biological processes, sleep is influenced by environmental, psychosocial, and cultural factors.

Understanding the relationship between parental factors and child sleep-wake patterns, alongside identifying potential developmental shifts during this period, is essential. However, existing research, often limited to cross-sectional or short-term longitudinal studies, has mostly focused on mothers, with few studies considering the transactional nature between infants' sleep patterns and the bidirectional influences exerted by other important parental factors.

This longitudinal study aims to understand how parent-infant interactions influence infant sleep patterns across the first three years of life for both mothers and fathers. The study will further examine the effects of parental factors, including (1) the co-parenting relationship, (2) maternal self-efficacy, (3) maternal/paternal depression, (4) maternal/paternal anxiety, (5) paternal involvement, (6) maternal/paternal sleep, and (7) parental stress, along with child factors such as temperament and socio-emotional development, on infants' sleep-wake patterns. Additionally, this study will investigate the dynamic, bidirectional relationships between these factors, providing valuable insights into infant and family well-being.

DETAILED DESCRIPTION:
Sleep is a physiological process for a child's healthy development, growth, and well-being. Although child sleep regulation across the early years proceeds well for many, estimates of sleep problems among infants range between 20-30%.

Beyond biological processes, sleep is influenced by environmental, psychosocial, and cultural factors. According to the transactional model, infant sleep is shaped through a bidirectional, continuous, and complex relationship between internal factors related to the infant (such as temperament) and factors related to the parents (such as parental mental health, sleep-related behaviors, and the quality of their relationship with the child). Cultural factors also play a significant role in shaping children's sleep patterns, influencing both their sleep habits and parents' approaches to addressing sleep issues. Understanding how parental factors and child sleep interact and evolve each other during the early years is vital for supporting the well-being of both infants and their families.

The primary objective of this study is to determine how parent-infant interactions influence changes in infant sleep patterns over the first three years of life, enabling the examination of bidirectional linkages and within-person associations between variations in parent and infant sleep. The second objective is to identify predictors of the relationship between parent and child sleep. Moreover, this study will enable the investigators to establish a birth cohort, which will serve as a valuable resource for addressing future research questions and advancing knowledge in this field.

This study adopts a longitudinal, prospective design. Families who are pregnant with first child in the second or third trimester will be invited to participate. Recruitment will take place from January to December 2025. Parents will be followed across seven time points: during pregnancy (second or third trimester) and at 3, 6, 12, 18, 24, and 36 months postpartum.

Sociodemographic information also will be collected. Parents will be assessed by Patient Health Questionnaire-9, Generalized Anxiety Disorder-7, Pittsburgh Sleep Quality Index, Coparenting Relationship Scale, Maternal Self-Efficacy Scale, Parental Stress Scale, Paternal Involvement Questionnaire. Sleep of children will be evaluated by the Turkish version of the expanded brief infant sleep questionnaire and the infant's social and emotional development will be assessed by Brief Infant Toddler Social Emotional Assessment. Child's temperament will be assessed with one question.

ELIGIBILITY:
Inclusion Criteria:

* Being pregnant with the first child Gestational age>12 weeks Parents over the age 18 Fluent in Turkish Parents living in Istanbul

Exclusion Criteria:

* Suicidal ideation in Patient Health Questionnaire-9 (PHQ-9) No internet access

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy pregnant women aged 18 and above and their partners
Sampling Method: Non-Probability Sample
Enrollment: 475 (Estimated)
Dates: Start 2025-01-21 (Actual); Primary Completion 2028-12-01 (Estimated); Study Completion 2028-12-01 (Estimated)

PRIMARY OUTCOMES:
Infant sleep-wake patterns | 3rd, 6th, 12th, 18th, 24th and 36th months
  Infant sleep wake patterns will be measured using the Revised-Brief Infant Sleep Questionnaire (BISQ-R). The BISQ-R is a parent-reported screening tool designed to evaluate sleep patterns in infants and young children. This scale consists of 33 questions with 19 questions for scoring. There are 3 subscales including infant sleep, parent perception and parent behavior. The total and each subscale score ranges from 0 to 100. Total score is the average of the 3 subscale scores. Higher scores indicate better sleep quality, more positive perception of infant sleep, and parental behaviors that promote healthy and independent sleep. The survey has been validated in Turkish.

SECONDARY OUTCOMES:
Prenatal co-parenting relationship | Baseline
  To evaluate prenatal coparenting relationships, the Coparenting Relationship Scale - Father's Prenatal Version will be used for both mother and fathers. The survey predicts that individuals with higher scores are more likely to have positive coparenting relationships in the future. The minimum score that can be obtained from the scale is 0, while the maximum score is 180.
Co-parenting relationship | 3rd, 6th, 12th, 18th, 24th and 36th months
  To evaluate coparenting relationships, the Coparenting Relationship Scale will be used which predicts that individuals with higher scores are more likely to have positive coparenting relationships. The minimum score that can be obtained from the scale is 0, while the maximum score is 150. The survey has been validated in Turkish.
Maternal Self Efficacy | 3rd, 6th, 12th, 18th, 24th and 36th months
  To evaluate maternal self efficacy, Maternal Self Efficacy Scale will be used. The survey is a ten item scale and a higher score on the scale indicates a higher level of maternal self-efficacy. The minimum score that can be obtained from the scale is 10, while the maximum score is 40. The survey has been validated in Turkish.
Maternal and Paternal Depression Symptoms | Baseline, 3rd, 6th, 12th, 18th, 24th and 36th months
  Parental depression symptoms will be measured with Patient Health Questionnaire-9. This nine-item scale is designed to assess the presence and severity of depressive symptoms. Based on the scale, scores of 0-4 indicate no depression, 5-9 indicate mild depression, and 10 or above reflect a high level of depression. The survey has been validated in Turkish.
Paternal Involvement | 12th. And 36th. months
  The Father Involvement Scale will be used to evaluate paternal involvement. This 37-item scale, scored using a 5-point Likert system, was developed for fathers with children aged 3 to 6 years. The survey assesses the frequency of one-on-one activities fathers engage in with their children and consists of three subscales: Playful Interaction, Basic Care, and Affection and Closeness. When the child is 12 months old, fathers will complete only the Basic Care and Affection and Closeness subscales, as these are more suitable for the child's age. At 36 months postpartum, fathers will be asked to complete the entire scale. Total scores range from a minimum of 37 to a maximum of 185, with higher scores indicating a greater level of paternal involvement.
Maternal and Paternal Sleep Quality | Baseline, 3rd, 6th, 12th, 18th, 24th and 36th months
  To evaluate maternal and paternal sleep, Pittsburgh Sleep Quality Index(PUKI) will be used. This survey is a 19-item self-report scale that evaluates sleep quality and disturbances over the past month. The total score ranges from 0 to 21. Higher scores on the scale are associated with lower sleep quality. The survey has been validated in Turkish.
Parental Stress | 3rd, 6th, 12th, 18th, 24th and 36th months
  To evaluate parental stress, the Parental Stress Scale will be used. This survey is a 16-item, 5-point Likert-type scale consisting of the subscales: Parental Rewards, Parental Stressors, Lack of Control, and Parental Satisfaction. In our study, only questions from the parental stressors subscale of the survey will be used. Higher scores indicate greater parental stress. The minimum score that can be obtained from the scale is 16, while the maximum score is 80. The survey has been validated in Turkish.
Child's Temperament | 3rd, 6th, 12th, 18th, 24th and 36th months
  Mothers and fathers will be asked to assess their baby's temperament with the question, "How would you evaluate your baby's temperament?" This will be rated on a 5-point Likert scale, with "1: Very easy" and "5: Very difficult."
Maternal and Paternal Anxiety | Baseline, 3rd, 6th, 12th, 18th, 24th and 36th months
  Maternal and paternal anxiety will be measured with Generalized Anxiety Scale-7. Scores on the scale are categorized as follows: 0-4 indicates mild anxiety, 5-9 moderate anxiety, 10-14 high anxiety, and 15-21 severe anxiety, with a cutoff score of 8 or higher. The survey has been validated in Turkish.
Infant's Social and Emotional Development | 12th., 18th., 24th. and 36th months
  Social and emotional development will be assessed using the Brief Infant Toddler Social Emotional Assessment (BITSEA), which comprises two domains: the Problem Scale, consisting of 31 items, and the Competence Scale, consisting of 11 items. Items are rated on a 3-point scale: 0 (not true/rarely), 1 (somewhat true/sometimes), and 2 (very true/often). The total score ranges from 0 to 62 for the Problem Scale and from 0 to 22 for the Competence Scale. Higher scores on the Problem Scale indicate a greater risk of emotional and behavioral problems, while lower scores on the Competence Scale suggest an increased risk of competence deficits or developmental delays. The survey has been validated in Turkish.

CONTACTS AND LOCATIONS:
Locations (1):
- Marmara University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided
Requests for wider sharing of data (for example in response to information on Marmara University webpages and in publications about the study and willingness to share), will be addressed on a case-by-case basis. Any data sharing request will be made to investigators through a pre-defined data requisition form. This form will contain information about the applicant, institution, purpose of data request, study objectives, ethical clearance of the study, etc. Once a request has been made the data governance body will discuss if that request was appropriate and meets the criteria set by the university; data will be released following signing of the data sharing agreement. The data will be stored on the Marmara University servers and not be deposited in any 'community' database.

REFERENCES:
- [Background] Karabekiroglu K, Rodopman-Arman A, Ay P, Ozkesen M, Akbas S, Tasdemir GN, Boke O, Peksen Y. The reliability and validity of the Turkish version of the brief infant-toddler social emotional assessment (BITSEA). Infant Behav Dev. 2009 Jun;32(3):291-7. doi: 10.1016/j.infbeh.2009.03.003. Epub 2009 May 2. PMID 19411111
- [Background] Williamson AA, Mindell JA, Hiscock H, Quach J. Longitudinal sleep problem trajectories are associated with multiple impairments in child well-being. J Child Psychol Psychiatry. 2020 Oct;61(10):1092-1103. doi: 10.1111/jcpp.13303. Epub 2020 Jul 26. PMID 32713013
- [Background] Teti DM, Gelfand DM. Behavioral competence among mothers of infants in the first year: the mediational role of maternal self-efficacy. Child Dev. 1991 Oct;62(5):918-29. doi: 10.1111/j.1467-8624.1991.tb01580.x. PMID 1756667
- [Background] Feinberg ME, Brown LD, Kan ML. A Multi-Domain Self-Report Measure of Coparenting. Parent Sci Pract. 2012 Jan 1;12(1):1-21. doi: 10.1080/15295192.2012.638870. Epub 2012 Jan 20. PMID 23166477
- [Background] Sadeh A. A brief screening questionnaire for infant sleep problems: validation and findings for an Internet sample. Pediatrics. 2004 Jun;113(6):e570-7. doi: 10.1542/peds.113.6.e570. PMID 15173539
- [Background] Buysse DJ, Reynolds CF 3rd, Monk TH, Berman SR, Kupfer DJ. The Pittsburgh Sleep Quality Index: a new instrument for psychiatric practice and research. Psychiatry Res. 1989 May;28(2):193-213. doi: 10.1016/0165-1781(89)90047-4. PMID 2748771
- [Background] Yazici Gulec M, Gulec H, Simsek G, Turhan M, Aydin Sunbul E. Psychometric properties of the Turkish version of the Patient Health Questionnaire-Somatic, Anxiety, and Depressive Symptoms. Compr Psychiatry. 2012 Jul;53(5):623-9. doi: 10.1016/j.comppsych.2011.08.002. Epub 2011 Oct 13. PMID 22000476
- [Background] Kroenke K, Spitzer RL, Williams JB. The PHQ-9: validity of a brief depression severity measure. J Gen Intern Med. 2001 Sep;16(9):606-13. doi: 10.1046/j.1525-1497.2001.016009606.x. PMID 11556941
- [Background] Spitzer RL, Kroenke K, Williams JB, Lowe B. A brief measure for assessing generalized anxiety disorder: the GAD-7. Arch Intern Med. 2006 May 22;166(10):1092-7. doi: 10.1001/archinte.166.10.1092. PMID 16717171
- [Background] Cook F, Conway LJ, Giallo R, Gartland D, Sciberras E, Brown S. Infant sleep and child mental health: a longitudinal investigation. Arch Dis Child. 2020 Jul;105(7):655-660. doi: 10.1136/archdischild-2019-318014. Epub 2020 Mar 9. PMID 32152038
- [Background] Boran P, Ergin A, Us MC, Dinleyici M, Velipasaoglu S, Yalcin SS, Barutcu A, Gokcay G, Gur E, Camurdan Duyan A, Aydin A, Celep G, Almis H, Savci G, Kondolot M, Nalbantoglu B, Unver Korgali E, Yendur O, Orhon Simsek F, Kara Uzun A, Bag O, Koc F, Bulbul S. Young children's sleep patterns and problems in paediatric primary healthcare settings: a multicentre cross-sectional study from a nationally representative sample. J Sleep Res. 2022 Dec;31(6):e13684. doi: 10.1111/jsr.13684. Epub 2022 Jul 5. PMID 35790464
- [Background] Sadeh A, Tikotzky L, Kahn M. Sleep in infancy and childhood: implications for emotional and behavioral difficulties in adolescence and beyond. Curr Opin Psychiatry. 2014 Nov;27(6):453-9. doi: 10.1097/YCO.0000000000000109. PMID 25247458
- [Background] Mindell JA, Sadeh A, Wiegand B, How TH, Goh DY. Cross-cultural differences in infant and toddler sleep. Sleep Med. 2010 Mar;11(3):274-80. doi: 10.1016/j.sleep.2009.04.012. Epub 2010 Feb 6. PMID 20138578
- [Background] Meltzer LJ, Williamson AA, Mindell JA. Pediatric sleep health: It matters, and so does how we define it. Sleep Med Rev. 2021 Jun;57:101425. doi: 10.1016/j.smrv.2021.101425. Epub 2021 Jan 19. PMID 33601324
- [Background] Covington LB, Patterson F, Hale LE, Teti DM, Cordova A, Mayberry S, Hauenstein EJ. The contributory role of the family context in early childhood sleep health: A systematic review. Sleep Health. 2021 Apr;7(2):254-265. doi: 10.1016/j.sleh.2020.11.010. Epub 2021 Jan 10. PMID 33436342